CLINICAL TRIAL: NCT03363204
Title: Interest of the BRUXENSE Occlusal Splints for Bruxism Diagnosis: a Feasibility Study
Acronym: BRUXENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0281
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bruxism, Sleep-Related
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRUXENSE (Experimental): Patients corresponding to selection criteria will use the BRUXENSE occlusal splint for 10 consecutive nights.
  Interventions: Device: BRUXENSE occlusal splint

INTERVENTIONS:
Device: BRUXENSE occlusal splint — Patients participating will put the BRUXENSE occlusal splint each night. During the night the device will collect data potentially related to bruxism. After each night the device will be cleaned with water and toothpaste and charged. This routine will be conducted over 10 consecutive nights.

SUMMARY:
There is no accurate diagnosis method for bruxism for now. Consequences of bruxism over teeth, muscles and articulation of the jaw are important.

This study aims to develop a innovative tool in order to accurately rapidly diagnose bruxism in ambulatory evaluation.

ELIGIBILITY:
Inclusion Criteria:

* adult from 18-70
* patients diagnosed with bruxism according to the following criteria:
* positive question at one of the following question:

  * are you aware of your grinding?
  * does your partner hear you grinding?
  * are you aware that you are frequently tighten your jaws during the day and/or the night?
  * are you tired and/or do experience jaws 'muscular pain in the morning.
* presence of at least one criteria:

  * abnormal tooth wear or tooth prosthesis damages
  * Hypertrophy of the masseter muscles
* patients agreeing to participate
* patient able to understand and follow the protocol
* patient with health insurance

Exclusion Criteria:

* patients with more than 2 missing tooth
* Severe troubles to correctly close the mouth.
* neurological disorder (Parkinson, Alzheimer) or psychiatric disorder
* Sleep disorder (insomnia, narcolepsy, sleep apnea, restless leg disorder)
* use of drugs that potentially impair sleep (benzodiazepines, neuroleptics, tricyclic antidepressants) alcohol or narcotics.
* complete or partial removal dental prosthesis or orthodontic device
* Patient under legal protection
* pregnant women
* Patients deprived of their freedom by a judicial or administrative decision

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Patient rate with successful use of BRUXENSE occlusal splint | At day 10
  The BRUXENSE occlusal splints correct use in real situation will be evaluated by measuring the percentage of subjects able to use this occlusal splints during 10 consecutive nights (6 hours minimum) without any pain or any discomfort. 10 nights is the necessary delay to record sufficient data to make a diagnosis.

SECONDARY OUTCOMES:
Number of usable measurements | At day 10
  The quality of collected data will be determined by the number of measurements that can be used to make a diagnosis of bruxism after 10 consecutive nights
Satisfaction scale score | At day 10
  Subject satisfaction will be assessed thanks to a numeric scale going from 0 (not satisfied at all) to 10 (completely satisfied)
Proportion of patients diagnosed with bruxism | At day 10
  Proportion of patients diagnosed with bruxism according to the BRUXENSE occlusal splints after the analysis of the data collected during 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Consultations et de Traitements Dentaires, Hospices Civils de Lyon, Lyon, France, France

REFERENCES:
- [Result] Robin O, Claude A, Gehin C, Massot B, McAdams E. Recording of bruxism events in sleeping humans at home with a smart instrumented splint. Cranio. 2022 Jan;40(1):14-22. doi: 10.1080/08869634.2019.1708608. Epub 2020 Jan 8. PMID 31914871